CLINICAL TRIAL: NCT02936453
Title: Efficacy of Spinal Epidural Electrical Stimulation (EES) in Combination With Robot-assisted Neurorehabilitation in Patients With Spinal Cord Injury (STIMO)
Brief Title: STIMO: Epidural Electrical Simulation (EES) With Robot-assisted Rehabilitation in Patients With Spinal Cord Injury.
Acronym: STIMO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jocelyne Bloch (Other)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (Other); Foundation Wings For Life (Other)
Responsible Party: Sponsor-Investigator, Jocelyne Bloch, Doctor, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STIMO2016
Record Dates: First submitted 2016-10-12; First posted 2016-10-18 (Estimated); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Epidural Electrical Stimulation; Robot-assisted
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): Patients will participate during 8-12 months, during which there will be :
  * Pre-implant evaluations (6-8 weeks)
  * Device implantation and stimulation optimization (6-8 weeks)
  * Overground rehabilitation training with EES (5-6 months) In the period after implantation participants need to be present at the CHUV University Hospital in Lausanne 4 days per week for testing and training (lodging can be provided). It is possible to complement the neuro-rehabilitative training at CHUV with a training outside the rehabilitation room by making use of the Home-use system.
  An optional extension of the study up to 3 years is offered. During this period, the patient can continue the training with the Home-use system.
  Interventions: Procedure: Device implantation

INTERVENTIONS:
Procedure: Device implantation — * Implantation of Specify 5-6-5 lead or Go-2 lead in epidural space
  * Implantation of Activa RC neurostimulator

SUMMARY:
STIMO is a First-in-Man (FIM) study to confirm the safety and feasibility of a closed-loop Epidural Electrical Stimulation (EES) in combination with overground robot assisted rehabilitation training for patients with chronic incomplete spinal cord injury (SCI).

Patients will participate during 8-12 months, during which there will be:

* Pre-implant evaluations (6-8 weeks)
* Device implantation and stimulation optimization (6-8 weeks)
* Overground rehabilitation training with EES (5-6 months). In the period after implantation, participants need to be present for testing and training, 4 days per week at the CHUV University Hospital in Lausanne (lodging can be provided). It is possible to complement the neuro-rehabilitative training at CHUV with training outside the rehabilitation room by making use of the Home-use system.

At the end of the protocol, the study aims to make the patients walk better and faster. As this is the first study of its kind, success is not guaranteed. However, the potential benefits outweigh the potential risks.

An optional extension of the study up to 3 years is offered. During this period, the patient can continue the training with the Home-use system.

DETAILED DESCRIPTION:
STIMO is a First-in-Man (FIM) study with the objective to confirm the safety and feasibility of a closed-loop Epidural Electrical Stimulation (EES) in combination with overground robot assisted rehabilitation training for patients with chronic incomplete spinal cord injury (SCI), as it was previously successfully demonstrated in animals.

The study consists of two phases:

A. Main study

The main study lasts about 8-12 months for each individual participant, from signing informed consent to the final test in the study This period can be divided into 3 distinct phases:

* Pre-implant : about 6-8 weeks from informed consent to implant. During this phase, patient will participate during a total of 6 distinct days of evaluations, of which 5 days in Lausanne and 1 day at the assessment center in Zurich. The patient will also participate to 3 weeks of pre-implantation training in a Body Weight Support (BWS) system.
* Implant and stimulation optimization: about 6-8 weeks, including the implantation of the epidural lead and the neurostimulator. In this phase, the optimal stimulation parameters will be determined for the flexing and stretching of both legs. During this period, participants need to be present at the CHUV University Hospital in Lausanne 4-5 days per week (lodging can be provided).
* Rehabilitation training and final evaluation: 4 days per week of rehabilitation training during a period of 5 months, followed by a final evaluation lasting 4 days in Lausanne and 1 day in Zurich. In this phase, the patients receive intensive overground rehabilitation training using a body weight support device in combination with EES, with the aim of significantly improving their walking capabilities. During this period, participants need to be present at the CHUV University Hospital in Lausanne (lodging can be provided) 4 days per week.

Once the patient has shown the ability to stand or walk safely without robotic assistance, he/she is offered the possibility to complement his/her neuro-rehabilitative training using EES outside the robotic environment and rehabilitation room by making use of the Home-use system.

B. Optional study extension (3 years)

The patient has the possibility to continue his/her neuro-rehabilitative training with the home-use system for an additional period of 3 years after the end of clinical rehabilitation period. During this period, evaluation measures and technical check-ups are made at regular time points. The patient is contacted monthly to ensure a normal training conduct and a safety follow-up.

At the end of the protocol, the study aims to make the patients walk better and faster. Improvements are quantified through pre-defined measures assessed prior to implant and at the end of the main study as well as at regular time points during the optional study extension.

As this is the first study of its kind, success is not guaranteed. However, the potential benefits outweigh the potential risks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 (women or men)
* Incomplete SCI graded as AIS A,B,C & D
* Level of lesion: T10 and above, based on AIS level determination by the PI, with preservation of conus function
* The intact distance between the cone and the lesion must be at least 60mm
* Focal spinal cord disorder caused by either trauma or epidural, subdural or intramedullary bleeding
* Minimum 12 months post-injury
* Completed in-patient rehabilitation program
* Able to stand with walker or 2 crutches
* Stable medical and physical condition as considered by Investigators
* Adequate care-giver support and access to appropriate medical care in patient's home community
* Agree to comply in good faith with all conditions of the study and to attend all required study training and visits
* Must participate in two training sessions before enrolment
* Must provide and sign Informed Consent prior to any study related procedures

Exclusion Criteria:

* Limitation of walking function based on accompanying (CNS) disorders (systemic malignant disorders, cardiovascular disorders restricting physical training, peripheral nerve disorders)
* History of significant autonomic dysreflexia
* Cognitive/brain damage
* Epilepsy
* Patient who has spinal canal stenosis
* Patient who uses an intrathecal Baclofen pump.
* Patient who has any active implanted cardiac device such as pacemaker or defibrillator.
* Patient who has any indication that would require diathermy.
* Patient who has any indication that would require MRI.
* Patient that have an increased risk for defibrillation
* Severe joint contractures disabling or restricting lower limb movements.
* Haematological disorders with increased risk for surgical interventions (increased risk of haemorrhagic events).
* Participation in another locomotor training study.
* Congenital or acquired lower limb abnormalities (affection of joints and bone).
* Women who are pregnant (pregnancy test obligatory for woman of childbearing potential) or breast feeding or not willing to take contraception.
* Known or suspected non-compliance, drug or alcohol abuse.
* Spinal cord lesion due to either a neurodegenerative disease or a tumour.
* Patient has other anatomic or co-morbid conditions that, in the investigator's opinion, could limit the patient's ability to participate in the study or to comply with follow-up requirements, or impact the scientific soundness of the study results.
* Patient is unlikely to survive the protocol follow-up period of 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Safety and Preliminary efficacy: Walking Index for Spinal Cord Injury (WISCI II) | 7 months after implant
  The Walking Index for Spinal Cord Injury is an ordinal scale that has been frequently used in clinical trials as a tool to assess walking function.
Safety and Preliminary efficacy: 10-Meter Walk Test (10MWT) | 7 months after implant
  10-Meter Walk Test (10MWT) is commonly used to measure walking speeds during two conditions: comfortable and fast. It yields scores that are valid and reliable for SCI individuals.
Safety and Preliminary efficacy: Weight Bearing Capacity (WBC). | 7 months after implant
  Weight-bearing capacity (WBC) is an important outcome to monitor and particularly relevant in patients with severe motor impairments who cannot walk independently.

SECONDARY OUTCOMES:
Improvement of walking capability: Spinal Cord Independence Measure (SCIM III). | 7 months after implant
  Spinal Cord Independence Measure (SCIM III) is a test used as a reference tool for the assessment of overall functional ability after SCI.
Improvement of walking capability: 6-Min Walk Test (6MWT). | 7 months after implant
  This assessment is a submaximal test that will be used as a global and easy indicator of the locomotor performance.

OTHER OUTCOMES:
ASIA Impairment Scale (AIS) | 7 months after implant
  The American Spinal Injury Association (ASIA) Standard Neurological Classification of Spinal Cord Injury is a standard method of assessing the neurological status, including motor and sensory evaluations, of a person who has sustained a spinal cord injury.
Modified Ashworth Scale (MAS) | 7 months after implant
  The Modified Ashworth Scale is a method for measuring muscle spasticity. It involves manual movement of a limb through its range of motion to passively stretch specific muscle groups.
Berg Balance Scale (BBS) | 7 months after implant
  The Berg Balance Scale was developed to measure balance among frail populations with impairment in balance function by assessing the performance of functional tasks with a 14-item scale.
Quality of life (pain, spasticity, bladder/bowel regulation, sex life and sleep) | 7 months after implant
  A dedicated set of questionnaires is selected to monitor the quality of life (QoL). The questionnaires are dedicated to the social participation to society as well as to the self-reported problems affecting the QoL of SCI individuals (pain, spasticity, bladder/bowel regulation, sex life and sleep).
Neurobiomechanical recordings | 7 months after implant
  Neurobiomechanical behaviour during different locomotor tasks will be recorded with a combination of kinematics, kinetics and EMG data.
Electrophysiological recordings and voluntary control of muscle contraction | 7 months after implant
  A dedicated set of tests is selected to assess a variety of physiological parameters.
Short Pain Assessment | 7 months after implant
  The pain assessment reports on the subjective feeling of pain during the previous week. It assesses the nature and location of pain and its interference with activities of daily living (ADL).

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire Courtine, Study Chair — Ecole Polytechnique Fédérale de Lausanne; Armin Curt, Study Chair — University Hospital Balgrist, Zuerich
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Angeli CA, Edgerton VR, Gerasimenko YP, Harkema SJ. Altering spinal cord excitability enables voluntary movements after chronic complete paralysis in humans. Brain. 2014 May;137(Pt 5):1394-409. doi: 10.1093/brain/awu038. Epub 2014 Apr 8. PMID 24713270
- [Background] Dominici N, Keller U, Vallery H, Friedli L, van den Brand R, Starkey ML, Musienko P, Riener R, Courtine G. Versatile robotic interface to evaluate, enable and train locomotion and balance after neuromotor disorders. Nat Med. 2012 Jul;18(7):1142-7. doi: 10.1038/nm.2845. PMID 22653117
- [Background] Harkema S, Gerasimenko Y, Hodes J, Burdick J, Angeli C, Chen Y, Ferreira C, Willhite A, Rejc E, Grossman RG, Edgerton VR. Effect of epidural stimulation of the lumbosacral spinal cord on voluntary movement, standing, and assisted stepping after motor complete paraplegia: a case study. Lancet. 2011 Jun 4;377(9781):1938-47. doi: 10.1016/S0140-6736(11)60547-3. Epub 2011 May 19. PMID 21601270
- [Background] van den Brand R, Heutschi J, Barraud Q, DiGiovanna J, Bartholdi K, Huerlimann M, Friedli L, Vollenweider I, Moraud EM, Duis S, Dominici N, Micera S, Musienko P, Courtine G. Restoring voluntary control of locomotion after paralyzing spinal cord injury. Science. 2012 Jun 1;336(6085):1182-5. doi: 10.1126/science.1217416. PMID 22654062
- [Background] Wenger N, Moraud EM, Raspopovic S, Bonizzato M, DiGiovanna J, Musienko P, Morari M, Micera S, Courtine G. Closed-loop neuromodulation of spinal sensorimotor circuits controls refined locomotion after complete spinal cord injury. Sci Transl Med. 2014 Sep 24;6(255):255ra133. doi: 10.1126/scitranslmed.3008325. PMID 25253676
- [Background] Wenger N, Moraud EM, Gandar J, Musienko P, Capogrosso M, Baud L, Le Goff CG, Barraud Q, Pavlova N, Dominici N, Minev IR, Asboth L, Hirsch A, Duis S, Kreider J, Mortera A, Haverbeck O, Kraus S, Schmitz F, DiGiovanna J, van den Brand R, Bloch J, Detemple P, Lacour SP, Bezard E, Micera S, Courtine G. Spatiotemporal neuromodulation therapies engaging muscle synergies improve motor control after spinal cord injury. Nat Med. 2016 Feb;22(2):138-45. doi: 10.1038/nm.4025. Epub 2016 Jan 18. PMID 26779815
- [Derived] Carroll AH, Fakhre E, Quinonez A, Tannous O, Mesfin A. An Update on Spinal Cord Injury and Current Management. JBJS Rev. 2024 Oct 24;12(10). doi: 10.2106/JBJS.RVW.24.00124. eCollection 2024 Oct 1. PMID 39446982
- [Derived] Rowald A, Komi S, Demesmaeker R, Baaklini E, Hernandez-Charpak SD, Paoles E, Montanaro H, Cassara A, Becce F, Lloyd B, Newton T, Ravier J, Kinany N, D'Ercole M, Paley A, Hankov N, Varescon C, McCracken L, Vat M, Caban M, Watrin A, Jacquet C, Bole-Feysot L, Harte C, Lorach H, Galvez A, Tschopp M, Herrmann N, Wacker M, Geernaert L, Fodor I, Radevich V, Van Den Keybus K, Eberle G, Pralong E, Roulet M, Ledoux JB, Fornari E, Mandija S, Mattera L, Martuzzi R, Nazarian B, Benkler S, Callegari S, Greiner N, Fuhrer B, Froeling M, Buse N, Denison T, Buschman R, Wende C, Ganty D, Bakker J, Delattre V, Lambert H, Minassian K, van den Berg CAT, Kavounoudias A, Micera S, Van De Ville D, Barraud Q, Kurt E, Kuster N, Neufeld E, Capogrosso M, Asboth L, Wagner FB, Bloch J, Courtine G. Activity-dependent spinal cord neuromodulation rapidly restores trunk and leg motor functions after complete paralysis. Nat Med. 2022 Feb;28(2):260-271. doi: 10.1038/s41591-021-01663-5. Epub 2022 Feb 7. PMID 35132264
- See also: Courtine-Lab is a part of the Center for Neuroprosthetic and Brain Mind Institute of the Life Science School at the Swiss Federal Institute of Technology Lausanne (EPFL). The laboratory is headed by Professor Grégoire Courtine. — http://courtine-lab.epfl.ch/